CLINICAL TRIAL: NCT03330457
Title: A Randomized, Double-blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenously Administered Andexanet After Dosing to Steady-State With Oral Betrixaban in Healthy Subjects
Brief Title: A Healthy Volunteer PK/PD, Safety and Tolerability Study of Andexanet After Betrixaban Dosing
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Ended prematurely
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-507
Record Dates: First submitted 2017-09-27; First posted 2017-11-06 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — PRT064445; betrixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Bertrixaban/Andexanet (Experimental): Andexanet 800 mg, administered as a slow IV bolus after having been dosed to steady-state with betrixaban 80 mg PO once daily (QD) for 7 days
  Interventions: Biological: Andexanet alfa (bolus); Drug: Betrixaban 80 mg PO QD
- Cohort 1 Bertrixaban/Placebo (Experimental): Placebo, administered as a slow IV bolus after having been dosed to steady-state with betrixaban 80 mg PO once daily (QD) for 7 days
  Interventions: Biological: Andexanet alfa (bolus); Drug: Betrixaban 80 mg PO QD; Biological: Andexanet alfa (infusion IV)
- Cohort 2 Bertrixaban/Andexanet (Experimental): andexanet 800 mg administered as a slow IV bolus at a target rate of approximately 30 mg/min followed by a continuous infusion of up to 8 mg/min for 120 min (960 mg) starting 4 h after the last dose of betrixaban
  Interventions: Biological: Andexanet alfa (bolus); Drug: Betrixaban 80 mg PO QD; Biological: Andexanet alfa (infusion IV)
- Cohort 2 Bertrixaban/Placebo (Experimental): Placebo administered as a slow IV bolus at a target rate of approximately 30 mg/min followed by a continuous infusion of up to 8 mg/min for 120 min (960 mg) starting 4 h after the last dose of betrixaban
  Interventions: Biological: Andexanet alfa (bolus); Drug: Betrixaban 80 mg PO QD; Biological: Andexanet alfa (infusion IV)

INTERVENTIONS:
Biological: Andexanet alfa (bolus) — fXa inhibitor antidote
Drug: Betrixaban 80 mg PO QD — fXa inhibitor
Biological: Andexanet alfa (infusion IV) — fXa inhibitor antidote
  Arms: Cohort 1 Bertrixaban/Placebo; Cohort 2 Bertrixaban/Andexanet; Cohort 2 Bertrixaban/Placebo

SUMMARY:
This is a randomized, double-blind, single center study in healthy volunteers dosed to steady state with betrixaban, designed to (1) Determine an andexanet dosing regimen required to reverse anticoagulant activity of betrixaban in healthy subjects, (2) Assess the safety and tolerability of andexanet vs. placebo (3) Determine the PK properties of andexanet and betrixaban (4) Determine the PD properties of betrixaban before, during, and after receiving andexanet or placebo and (5) Investigate the immunogenicity of andexanet in the presence of betrixaban.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a healthy man or woman between the ages of 18 and 45 years old, inclusive, who agrees to comply with the contraception and reproduction restrictions of the study:

   Men must be using two acceptable methods of contraception, at least one of which must be a barrier method (e.g., spermicidal gel plus condom) for the entire duration of the study and for at least three months following last study drug administration, and refrain from attempting to father a child or donating sperm in the three (3) months following the last study drug administration. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

   OR Men who report surgical sterilization (e.g., bilateral vasectomy) must have had the procedure at least six (6) months prior to initial dosing. Surgical sterilization procedures should be supported with clinical documentation and noted in the Relevant Medical History/Current Medical Conditions section of the Case report forms (CRFs).

   Women of childbearing potential must be using two medically acceptable methods of contraception, at least one of which must be a barrier method, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.), from the time of screening and for the duration of the study, through at least three months following last study drug administration. NOTE: Oral contraceptive use is not permitted due to their increased risk of thromboembolism. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

   OR Postmenopausal women must have had no regular menstrual bleeding for at least one (1) year prior to initial dosing. Menopause will be confirmed by an elevated plasma Follicle-stimulating hormone (FSH) level > 40mIU/mL at screening for women not in receipt of hormone replacement therapy (HRT); OR Women who report surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy) must have had the procedure at least six (6) months prior to initial dosing. Surgical sterilization procedures should be supported with clinical documentation and noted in the Relevant Medical History/Current Medical Conditions section of the CRF.

   AND All women must have a documented negative pregnancy test result at screening and at baseline.
2. The subject has clinically unremarkable medical history, physical examination, ECG, and vital signs, as determined by the Investigator. Laboratory values must also be clinically unremarkable as determined by the Investigator, with the exception of the following labs which must be strictly within the normal range:

   1. Coagulation labs - PT, aPTT, ACT;
   2. Hematology lab - Hematocrit/Hemoglobin;
   3. Liver function labs - Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) (may be below lower limit of normal [LLN], but not above upper limit of normal [ULN]).
3. The subject has a body mass index 19 to 30 kg/m2, inclusive, and weighs at least 60 kg.
4. The subject agrees to abstain from alcohol consumption for 48 hours prior to dosing and for the duration of the in-house study period.
5. The subject smokes <4 cigarettes/day (or equivalent: ≤0.5 can of chewing tobacco/week, 1 cigar/day) and agrees to abstain from smoking while domiciled.
6. The subject is able to read and give written informed consent and has signed a consent form approved by the Investigator's Institutional Review Board (IRB) or Ethics Committee (EC).

Exclusion Criteria:

1. The subject has a known history (including family history) of, symptoms of, or risk factors for bleeding (e.g., prior gastrointestinal bleeding, known berry aneurysm/ vascular malformation) or a stool specimen within 6 months of randomization that is positive for occult blood.
2. The subject has an absolute/relative contraindication to anticoagulation.
3. The subject has a history (including family history) of or risk factors for a hypercoagulable or thrombotic condition (e.g., deep vein thrombosis/pulmonary embolism, Factor V Leiden carrier).
4. The subject has a history of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease or condition which is known to make the subject susceptible to volume overload.
5. The subject has taken any prescription drugs (including oral contraceptives/HRT) or illicit drugs in the 30 days prior to randomization. The subject is also excluded if he/she has taken over the counter drugs, including dietary supplements and herbal products, in the 2 weeks prior to randomization. Furthermore, the subject agrees not to take any such drugs throughout the study (if it becomes medically necessary to do so, the Investigator and Portola Medical Monitor must be informed immediately).
6. The subject has a history of major surgery, severe trauma or bone fracture within 3 months prior to dosing; or planned surgery within 1 month after dosing.
7. The subject has a history of blood donation of more than 500 mL within 3 months prior to dosing.
8. The subject has participated in an investigational drug study within 30 days or 5 half-lives of the investigational compound, whichever is greater, of Day -1.
9. The subject has a positive screen for drugs of abuse at Day -1.
10. The subject has a medical or surgical condition which may impair drug absorption.
11. The subject is allergic to any of the vehicle ingredients: tris, arginine, hydrochloric acid, sucrose and polysorbate 80.
12. Subject is breastfeeding.
13. The subject has any condition which could interfere with or for which the treatment might interfere with the conduct of the study, or which would, in the opinion of the Investigator increase the risk of the subject's participation in the study. This would include, but is not limited to alcoholism, drug dependency or abuse, psychiatric disease, epilepsy or any unexplained blackouts.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: healthy subjects
Pre-assignment Details: 18 subjects met the inclusion/exclusion criteria; 18 subjects were randomized to two cohorts (6 andexanet and 3 placebo each cohort)
Period: Overall Study
Arm/Group | Cohort 1 Bertrixaban/Andexanet | Cohort 1 Bertrixaban/Placebo | Cohort 2 Bertrixaban/Andexanet | Cohort 2 Bertrixaban/Placebo
Started | 6 | 3 | 6 | 3
Completed | 6 | 3 | 6 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population will consist of all subjects randomized and treated with at least one dose of study medication (andexanet, andexanet placebo, or betrixaban). All safety analyses will be performed by actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Bertrixaban/Andexanet | Cohort 1 Bertrixaban/Placebo | Cohort 2 Bertrixaban/Andexanet | Cohort 2 Bertrixaban/Placebo | Total
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (3.6) | 37.3 (10.8) | 30.0 (3.7) | 36.3 (10.8) | 35.1 (7.0)
Age, Continuous [Median (Full Range); unit: years] | 39.5 [33.0 to 42.0] | 42.0 [25.0 to 45.0] | 31.0 [25.0 to 34.0] | 41.0 [24.0 to 44.0] | 34.5 [24.0 to 45.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 2 | 9
  Male | 2 | 2 | 4 | 1 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Anti-Fxa Activity From Baseline to End of Bolus
Description: Change in Anti-Fxa Activity from baseline to end of bolus
Time Frame: Baseline to end of bolus, approximately 2.5 hours
Population: The PD analysis populations will consist of all subjects who have received the requisite treatments and have data at any required time points.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Cohort 1 Bertrixaban/Andexanet | Cohort 1 Bertrixaban/Placebo | Cohort 2 Bertrixaban/Andexanet | Cohort 2 Bertrixaban/Placebo
Number analyzed (Participants) | 6 | 3 | 6 | 3
ug/L | -23.45 (7.453) | -1.67 (10.090) | -26.17 (16.661) | -2.17 (4.065)

2. Secondary Outcome: Change in Thrombin Generation From Baseline to End of Bolus
Description: Change in Thrombin Generation from baseline to end of bolus
Time Frame: Baseline to end of bolus, approximately 2.5 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: RFU
Arm/Group | Cohort 1 Bertrixaban/Andexanet | Cohort 1 Bertrixaban/Placebo | Cohort 2 Bertrixaban/Andexanet | Cohort 2 Bertrixaban/Placebo
Number analyzed (Participants) | 6 | 3 | 6 | 3
RFU | 129984.5 (39858.49) | 28646.7 (43991.66) | 116834.7 (49006.72) | 15998.7 (18081.07)

ADVERSE EVENTS:
Time Frame: Study day 1 to 48(+3)
Description: AEs, both serious and non-serious, occurring between signing informed consent and through the Termination Visit will be recorded on the eCRFs. All AEs/SAEs should be monitored until they are resolved, are not expected to improve further, or are determined to be due to a stable or chronic condition or intercurrent illness. Any AE/SAE that occurs with an onset date > 30 days after study completion and that the Investigator considers to be related to study medication, must be reported to Portola.
Arm/Group | Cohort 1 Bertrixaban/Andexanet | Cohort 1 Bertrixaban/Placebo | Cohort 2 Bertrixaban/Andexanet | Cohort 2 Bertrixaban/Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 1/6 | 0/3 | 2/6 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Bertrixaban/Andexanet (N=6) | Cohort 1 Bertrixaban/Placebo (N=3) | Cohort 2 Bertrixaban/Andexanet (N=6) | Cohort 2 Bertrixaban/Placebo (N=3)
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vessel Puncture Site Haemorrhage (General disorders) | 1 | 0 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes